CLINICAL TRIAL: NCT01084239
Title: Rule Out Myocardial Ischemia/Infarction by Computer Assisted Tomography
Brief Title: Multicenter Study to Rule Out Myocardial Infarction by Cardiac Computed Tomography
Acronym: ROMICAT-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Kaiser Permanente (Other); Beth Israel Deaconess Medical Center (Other); Bay State Clinical Trials, Inc. (Other); Washington University School of Medicine (Other); Tufts Medical Center (Other); The Cleveland Clinic (Other); Northwestern University (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Udo Hoffmann, MD MPH, Director of Cardiac Imaging, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009P002331
Record Dates: First submitted 2010-01-07; First posted 2010-03-10 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina Pectoris
Keywords: acute chest pain; emergency department; cardiac computed tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (No Intervention): Subjects in this arm (50% of the total cohort) continued to receive standard non-invasive evaluation of acute chest pain symptoms in the emergency department - mostly comprising of, but not limited to - exercise treadmill test, stress test with imaging and stress echocardiography.
- Cardiac CT (Experimental): Subjects in this arm (50% of the total cohort) were randomized to receive a cardiac computed tomography scan as part of the initial evaluation of acute chest pain symptoms, upon presentation to the emergency department.
  Interventions: Radiation: Cardiac Computed Tomography

INTERVENTIONS:
Radiation: Cardiac Computed Tomography — A contrast enhanced cardiac CT was performed in addition to standard evaluation. Reconstructed data sets were evaluated for the presence of coronary artery calcium, coronary atherosclerotic plaque and stenosis, LV function and incidental findings.
  Arms: Cardiac CT

SUMMARY:
The growing availability of cardiac computed tomography (CT)* in emergency departments (EDs) across the U.S. expands the opportunities for its clinical application, but also heightens the need to define its appropriate use in the evaluation of patients with acute chest pain. To address this need, we performed a randomized diagnostic trial (RDT) to determine whether integrating cardiac CT, along with the information it provides on coronary artery disease (CAD) and left ventricular (LV) function, can improve the efficiency of the management of these patients (i.e. shorten length of hospital stay, increase direct discharge rates from the ED, decreasing healthcare costs and improving cost effectiveness while being safe).

DETAILED DESCRIPTION:
Patients with acute chest pain and normal or non-diagnostic electrocardiograms (ECGs) represent a cohort whose management is notably inefficient and diagnostically challenging. Because in less than 30% of EDs diagnostic testing (e.g. nuclear imaging, echocardiography, and exercise treadmill ECG) that would allow physicians to rule out the occurrence of myocardial ischemia is performed as part of the initial evaluation, most of these patients are hospitalized for 24 to 36 hours to exclude the presence of acute coronary syndrome (ACS). Of the six million acute chest pain patients admitted each year in the U.S. under these conditions, less than 10% of them ultimately receive a diagnosis of ACS at discharge. Moreover, inpatient care for negative evaluations imparts an economic burden in excess of $8 billion annually.

Since acute myocardial ischemia and necrosis are rare in the absence of coronary artery disease, a technology that reliably identifies CAD may allow physicians to discharge chest pain patients directly from the ED. Cardiac CT is a safe, high-speed, noninvasive imaging technique that accurately detects coronary atherosclerotic plaque and stenosis, and also allows physicians to assess global and regional LV function.

Observational studies have demonstrated that approximately 40% of acute chest pain patients have no evidence of atherosclerosis on cardiac CT, and that an additional 30% have no evidence of hemodynamically significant (>50%) coronary artery stenosis. Both of these criteria are powerful predictors of the absence of both ACS and major adverse cardiovascular events (negative predictive value [NPV] of 98%). The specificity of cardiac CT is further increased when global and regional LV function is normal. Several studies have demonstrated that cardiac CT, with its high NPV, can be effectively used to rule out ACS, but little is known about the willingness ability of ED physicians to use this information to augment patient management.

We therefore performed a trial at 9 clinical sites and randomized 1000 patients with acute chest pain and normal or non-diagnostic ECGs, to receive either standard ED evaluation (no intervention) or a cardiac CT (experimental) in the evaluation of acute chest pain in the emergency room. (Rule Out Myocardial Infarction using Computer Assisted Computed Tomography [ROMICAT II]).

ELIGIBILITY:
Inclusion Criteria:

1. Participant had at least five minutes of chest pain or equivalent (chest tightness; pain radiating to left, right, or both arms or shoulders, back, neck, epigastrium, jaw/throat; or unexplained shortness of breath, syncope/presyncope, generalized weakness, nausea, or vomiting thought to be of cardiac origin) at rest or during exercise within 24 hours of ED presentation, warranting further risk stratification, as determined by an ED attending.
2. 2 or more cardiac risk factors (diabetes, hypertension, hyperlipidemia, current smoker and family history of coronary artery disease).
3. Able to provide a written informed consent.
4. <75 years of age, but >40 years of age.
5. Able to hold breath for at least 10 seconds.
6. Sinus rhythm.

Exclusion Criteria:

1. New diagnostic ischemic ECG changes (ST-segment elevation or depression > 1 mm or T-wave inversion > 4 mm) in more than two anatomically adjacent leads or left bundle branch block
2. Documented or self-reported history of CAD (MI, percutaneous coronary interventions [PCIs], coronary artery bypass graft [CABG], known significant coronary stenosis [>50%])
3. Greater than 6 hours since presentation to ED.
4. BMI >40 kg/m2
5. Impaired renal function as defined by serum creatinine >1.5 mg/dL*
6. Elevated troponin-T (> 0.09 ng/ml)
7. Hemodynamically or clinically unstable condition (BP systolic < 80 mm Hg, atrial or ventricular arrhythmias, persistent chest pain despite adequate therapy)
8. Known allergy to iodinated contrast agent
9. Currently symptomatic asthma
10. Documented or self-reported cocaine use within the past 48 hours (acute)
11. On Metformin therapy and unable or unwilling to discontinue for 48 hours after the CT scan
12. Contraindication to beta blockers (taking daily antiasthmatic medication): This exclusion only applies to patients with a heart rate >65 bpm at sites using a non-dual source CT scanner
13. Participant with no telephone or cell phone numbers or no address (preventing follow-up)
14. Participant with positive pregnancy test. Women of childbearing potential, defined as <2 years of menopause in the absence of hysterectomy or tube ligation, must have a pregnancy test performed within 24 hours before the CT scan.
15. Participant unwilling to provide a written informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Hoffmann, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Karady J, Mayrhofer T, Januzzi JL, Udelson JE, Fleg JL, Merkely B, Lu MT, Peacock WF, Nagurney JT, Koenig W, Ferencik M, Hoffmann U. Agreement among high-sensitivity cardiac troponin assays and non-invasive testing, clinical outcomes, and quality-of-care outcomes based on the 2020 European Society of Cardiology Guidelines. Eur Heart J Acute Cardiovasc Care. 2024 Feb 9;13(1):15-23. doi: 10.1093/ehjacc/zuad146. PMID 38001050
- [Derived] Karady J, Mayrhofer T, Ferencik M, Nagurney JT, Udelson JE, Kammerlander AA, Fleg JL, Peacock WF, Januzzi JL Jr, Koenig W, Hoffmann U. Discordance of High-Sensitivity Troponin Assays in Patients With Suspected Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Mar 30;77(12):1487-1499. doi: 10.1016/j.jacc.2021.01.046. PMID 33766254
- [Derived] Reinhardt SW, Babatunde A, Novak E, Brown DL. Effect of Race on Outcomes Following Early Coronary Computed Tomographic Angiography or Standard Emergency Department Evaluation for Acute Chest Pain. Ethn Dis. 2018 Oct 18;28(4):517-524. doi: 10.18865/ed.28.4.517. eCollection 2018 Fall. PMID 30405295
- [Derived] Bittner DO, Mayrhofer T, Puchner SB, Lu MT, Maurovich-Horvat P, Ghemigian K, Kitslaar PH, Broersen A, Bamberg F, Truong QA, Schlett CL, Hoffmann U, Ferencik M. Coronary Computed Tomography Angiography-Specific Definitions of High-Risk Plaque Features Improve Detection of Acute Coronary Syndrome. Circ Cardiovasc Imaging. 2018 Aug;11(8):e007657. doi: 10.1161/CIRCIMAGING.118.007657. PMID 30354493
- [Derived] Reinhardt SW, Lin CJ, Novak E, Brown DL. Noninvasive Cardiac Testing vs Clinical Evaluation Alone in Acute Chest Pain: A Secondary Analysis of the ROMICAT-II Randomized Clinical Trial. JAMA Intern Med. 2018 Feb 1;178(2):212-219. doi: 10.1001/jamainternmed.2017.7360. PMID 29138794
- [Derived] Ferencik M, Mayrhofer T, Lu MT, Woodard PK, Truong QA, Peacock WF, Bamberg F, Sun BC, Fleg JL, Nagurney JT, Udelson JE, Koenig W, Januzzi JL, Hoffmann U. High-Sensitivity Cardiac Troponin I as a Gatekeeper for Coronary Computed Tomography Angiography and Stress Testing in Patients with Acute Chest Pain. Clin Chem. 2017 Nov;63(11):1724-1733. doi: 10.1373/clinchem.2017.275552. Epub 2017 Sep 18. PMID 28923845
- [Derived] Bittner DO, Mayrhofer T, Bamberg F, Hallett TR, Janjua S, Addison D, Nagurney JT, Udelson JE, Lu MT, Truong QA, Woodard PK, Hollander JE, Miller C, Chang AM, Singh H, Litt H, Hoffmann U, Ferencik M. Impact of Coronary Calcification on Clinical Management in Patients With Acute Chest Pain. Circ Cardiovasc Imaging. 2017 May;10(5):e005893. doi: 10.1161/CIRCIMAGING.116.005893. PMID 28487318
- [Derived] Truong QA, Schulman-Marcus J, Zakroysky P, Chou ET, Nagurney JT, Fleg JL, Schoenfeld DA, Udelson JE, Hoffmann U, Woodard PK. Coronary CT Angiography Versus Standard Emergency Department Evaluation for Acute Chest Pain and Diabetic Patients: Is There Benefit With Early Coronary CT Angiography? Results of the Randomized Comparative Effectiveness ROMICAT II Trial. J Am Heart Assoc. 2016 Mar 22;5(3):e003137. doi: 10.1161/JAHA.115.003137. PMID 27006119
- [Derived] Pursnani A, Celeng C, Schlett CL, Mayrhofer T, Zakroysky P, Lee H, Ferencik M, Fleg JL, Bamberg F, Wiviott SD, Truong QA, Udelson JE, Nagurney JT, Hoffmann U. Use of Coronary Computed Tomographic Angiography Findings to Modify Statin and Aspirin Prescription in Patients With Acute Chest Pain. Am J Cardiol. 2016 Feb 1;117(3):319-24. doi: 10.1016/j.amjcard.2015.10.052. Epub 2015 Nov 18. PMID 26762723
- [Derived] Ferencik M, Liu T, Mayrhofer T, Puchner SB, Lu MT, Maurovich-Horvat P, Pope JH, Truong QA, Udelson JE, Peacock WF, White CS, Woodard PK, Fleg JL, Nagurney JT, Januzzi JL, Hoffmann U. hs-Troponin I Followed by CT Angiography Improves Acute Coronary Syndrome Risk Stratification Accuracy and Work-Up in Acute Chest Pain Patients: Results From ROMICAT II Trial. JACC Cardiovasc Imaging. 2015 Nov;8(11):1272-1281. doi: 10.1016/j.jcmg.2015.06.016. Epub 2015 Oct 14. PMID 26476506
- [Derived] Januzzi JL, Sharma U, Zakroysky P, Truong QA, Woodard PK, Pope JH, Hauser T, Mayrhofer T, Nagurney JT, Schoenfeld D, Peacock WF, Fleg JL, Wiviott S, Pang PS, Udelson J, Hoffmann U. Sensitive troponin assays in patients with suspected acute coronary syndrome: Results from the multicenter rule out myocardial infarction using computer assisted tomography II trial. Am Heart J. 2015 Apr;169(4):572-8.e1. doi: 10.1016/j.ahj.2014.12.023. Epub 2015 Jan 9. PMID 25819865
- [Derived] Pursnani A, Chou ET, Zakroysky P, Deano RC, Mamuya WS, Woodard PK, Nagurney JT, Fleg JL, Lee H, Schoenfeld D, Udelson JE, Hoffmann U, Truong QA. Use of coronary artery calcium scanning beyond coronary computed tomographic angiography in the emergency department evaluation for acute chest pain: the ROMICAT II trial. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002225. doi: 10.1161/CIRCIMAGING.114.002225. Epub 2015 Feb 20. PMID 25710925
- [Derived] Puchner SB, Liu T, Mayrhofer T, Truong QA, Lee H, Fleg JL, Nagurney JT, Udelson JE, Hoffmann U, Ferencik M. High-risk plaque detected on coronary CT angiography predicts acute coronary syndromes independent of significant stenosis in acute chest pain: results from the ROMICAT-II trial. J Am Coll Cardiol. 2014 Aug 19;64(7):684-92. doi: 10.1016/j.jacc.2014.05.039. PMID 25125300
- [Derived] Truong QA, Hayden D, Woodard PK, Kirby R, Chou ET, Nagurney JT, Wiviott SD, Fleg JL, Schoenfeld DA, Udelson JE, Hoffmann U. Sex differences in the effectiveness of early coronary computed tomographic angiography compared with standard emergency department evaluation for acute chest pain: the rule-out myocardial infarction with Computer-Assisted Tomography (ROMICAT)-II Trial. Circulation. 2013 Jun 25;127(25):2494-502. doi: 10.1161/CIRCULATIONAHA.113.001736. Epub 2013 May 17. PMID 23685743
- [Derived] Hoffmann U, Truong QA, Schoenfeld DA, Chou ET, Woodard PK, Nagurney JT, Pope JH, Hauser TH, White CS, Weiner SG, Kalanjian S, Mullins ME, Mikati I, Peacock WF, Zakroysky P, Hayden D, Goehler A, Lee H, Gazelle GS, Wiviott SD, Fleg JL, Udelson JE; ROMICAT-II Investigators. Coronary CT angiography versus standard evaluation in acute chest pain. N Engl J Med. 2012 Jul 26;367(4):299-308. doi: 10.1056/NEJMoa1201161. PMID 22830462
- [Derived] Hoffmann U, Truong QA, Fleg JL, Goehler A, Gazelle S, Wiviott S, Lee H, Udelson JE, Schoenfeld D; ROMICAT II. Design of the Rule Out Myocardial Ischemia/Infarction Using Computer Assisted Tomography: a multicenter randomized comparative effectiveness trial of cardiac computed tomography versus alternative triage strategies in patients with acute chest pain in the emergency department. Am Heart J. 2012 Mar;163(3):330-8, 338.e1. doi: 10.1016/j.ahj.2012.01.028. Epub 2012 Feb 22. PMID 22424002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment began on April 23, 2010, and ended on January 30, 2012, at nine hospitals in the United States.
Groups:
- Cardiac CT: Subjects in this arm (50% of the total cohort) were randomized to receive a cardiac computed tomography scan as part of the initial evaluation of acute chest pain symptoms, upon presentation to the emergency department.
  Cardiac Computed Tomography : A contrast enhanced cardiac CT was performed in addition to standard evaluation. Reconstructed data sets were evaluated for the presence of coronary artery calcium, coronary atherosclerotic plaque and stenosis, LV function and incidental findings.
Period: Randomization - Index Hospitalization
Arm/Group | Cardiac CT | Standard of Care
Started | 501 | 499
Completed | 501 | 499
Not Completed | 0 | 0
Period: 28-Day Follow-up
Arm/Group | Cardiac CT | Standard of Care
Started | 501 (All 501 patients enrolled were evaluated for follow-up at 28 days.) | 499
Completed | 497 | 490
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac CT | Standard of Care | Total
Number analyzed (Participants) | 501 | 499 | 1000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 433 | 440 | 873
  >=65 years | 68 | 59 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8) | 54 (8) | 54 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 229 | 468
  Male | 262 | 270 | 532
Region of Enrollment [Number; unit: participants]
  United States | 501 | 499 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Time Frame: Duration of stay in the hospital during the initial visit
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Cardiac CT: Subjects in this arm (50% of the total cohort) will be randomized to receive a cardiac computed tomography scan as part of the initial evaluation of acute chest pain symptoms, upon presentation to the emergency department.
  Cardiac Computed Tomography : A contrast enhanced cardiac CT will be performed in addition to standard evaluation. Reconstructed data sets will be evaluated for the presence of coronary artery calcium, coronary atherosclerotic plaque and stenosis, LV function and incidental findings.
- Standard of Care: Subjects in this arm (50% of the total cohort) will continue to receive standard non-invasive evaluation of acute chest pain symptoms in the emergency department - mostly comprising of, but not limited to - exercise treadmill test, stress test with imaging and stress echocardiography.
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
hours | 23.2 (37.0) | 30.8 (28.0)

2. Secondary Outcome: Time to Diagnosis
Time Frame: Time from ED arrival to first positive test (all tests except Echocardiography Rest and including troponins ) if discharge diagnosis is ACS, otherwise time to performance of last test (all tests except Echocardiography Rest and including troponins ).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
hours | 10.4 (12.6) | 18.7 (11.8)

3. Secondary Outcome: Healthcare Utilization
Description: Number of patients with diagnostic testing (CCTA, ETT, SPECT, stress echocardiography, and invasive coronary angiography)
Time Frame: Duration of stay in the hospital during the initial visit
Measure: Number; unit: participants
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
participants | 492 | 390
Statistical Analysis 1: Comparison: Cardiac CT vs Standard of Care; Test type: Superiority or Other; p < 0.001, Fisher Exact; Result for index hospitalization

4. Secondary Outcome: MACE
Description: Major Adverse Cardiovascular Events, All though these events are called MACE they do not qualify as adverse or serious adverse events. As these events are expected in some individuals in this population. Only MACE that occured within 72 hours after hospital discharge were considered serious adverse events in this trial. There were no such events.
Time Frame: 72 hours after discharge up to 28 days after enrollment.
Measure: Number; unit: events
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
events | 6 | 2

5. Secondary Outcome: Cost-effectiveness
Description: Total cost during index hospitalization
Time Frame: Duration of stay in the hospital during the initial visit
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
US Dollars | 4026 (6792) | 3874 (5298)

6. Secondary Outcome: Rate of ED Discharge
Description: Direct discharge from Emergency Department
Time Frame: Duration of stay in the hospital during the initial visit
Measure: Number; unit: participants
Arm/Group | Cardiac CT | Standard of Care
Number analyzed (Participants) | 501 | 499
participants | 233 | 62

ADVERSE EVENTS:
Arm/Group | Cardiac CT | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/501 | 0/499
Other Adverse Events (participants affected / at risk) | 5/501 | 1/499
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac CT (N=501) | Standard of Care (N=499)
Nausea and vomiting (General disorders) | 1 (1) | 0 (0) — one episode N/V after CTA contrast. Pt given 4mg zofran IV, symptoms resolved.
Nausea (General disorders) | 1 (1) | 0 (0) — Patient developed nausea immediately after administration of IV contrast, she has had IV contrast in the past without associated nausea.
RASH URTICARIAL (Eye disorders) | 1 (1) | 0 (0) — The patient developed a mild urticarial rash (2 separate quarter sized patches, 1 superior-lateral to his right eye and 1 superior-medial to his left eye) and associated itchiness within minutes of the injection of IV contrast.
ALLERGIC REACTION (General disorders) | 2 (2) | 0 (0)
THROMBOSIS ARTERIAL (General disorders) | 0 (0) | 1 (1) — right groin pseudoaneurysm

LIMITATIONS AND CAVEATS:
Enrollment occurred only during weekday hours.

Lack of blinding to the intervention.

Results may not be applicable to populations we did not study (i.e. patients younger than 40 years of age and those older than 74 years of age).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No